CLINICAL TRIAL: NCT02518113
Title: A Phase 1b/Randomized Phase 2 Study to Evaluate LY3039478 in Combination With Dexamethasone in T-ALL/T-LBL Patients
Brief Title: A Study of LY3039478 in Combination With Dexamethasone in Participants With T-ALL/T-LBL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14548; I6F-MC-JJCB (Other: Eli Lilly and Company); 2014-005024-10 (EudraCT Number)
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; T-cell Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — crenigacestat; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY3039478 + Dexamethasone (Adult) (Experimental): Part A: 50 mg LY3039478 administered orally three times per week (TIW) and 24 mg dexamethasone administered orally on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
  75 mg LY3039478 administered orally three times per week (TIW) and 24 mg dexamethasone administered orally on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
  100 mg LY3039478 administered orally three times per week (TIW) and 24 mg dexamethasone administered orally on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
  125 mg LY3039478 administered orally three times per week (TIW) and 24 mg dexamethasone administered orally on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
  Interventions: Drug: LY3039478; Drug: Dexamethasone
- LY3039478 + Dexamethasone (Pediatric) (Experimental): Part B: LY3039478 administered orally TIW at escalating doses and dexamethasone administered orally twice a day (BID) on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
  There were no participants enrolled to Part B of the study.
  Interventions: Drug: LY3039478; Drug: Dexamethasone
- Phase 2: LY3039478 + Dexamethasone (Experimental): LY3039478 administered orally TIW and dexamethasone administered orally BID on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
  There were no participants enrolled to Phase 2 of the study.
  Interventions: Drug: LY3039478; Drug: Dexamethasone
- Phase 2: Placebo + Dexamethasone (Placebo Comparator): Placebo administered orally TIW and dexamethasone administered orally BID on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
  There were no participants enrolled to Phase 2 of the study.
  Interventions: Drug: Dexamethasone; Drug: Placebo

INTERVENTIONS:
Drug: LY3039478 — Administered orally
  Arms: LY3039478 + Dexamethasone (Adult); LY3039478 + Dexamethasone (Pediatric); Phase 2: LY3039478 + Dexamethasone
Drug: Dexamethasone — Administered orally
Drug: Placebo — Administered orally
  Arms: Phase 2: Placebo + Dexamethasone

SUMMARY:
The main purpose of this study is to evaluate the safety of the study drug known as LY3039478 in combination with dexamethasone in participants with T-cell acute lymphoblastic leukemia or T-cell lymphoblastic lymphoma (T-ALL/T-LBL).

ELIGIBILITY:
Inclusion Criteria:

* Have acute T-cell lymphoblastic leukemia (T-ALL) or T-cell lymphoblastic lymphoma (T-LBL).
* T-ALL or T-LBL participants with relapsed/refractory disease.
* Have had at least 60 days between prior hematopoietic stem cell transplantation (SCT) and first dose of study drug.
* Have a performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) scale for adults.
* Lansky score >50% for participants <16 years old.
* Have adequate organ function.
* Are at least:

  * adult Phase 1 Part A and Phase 2: ≥16 years old at the time of screening
  * pediatric Phase 1 Part B: 2 to <16 years old
* Men and women with reproductive potential: Must agree to use a reliable method of birth control during the study and for 3 months following the last dose of study drug(s) or country requirements, whichever is longer.
* Females with childbearing potential: Have had a negative serum pregnancy test ≤7 days before the first dose of study drug and also must not be breastfeeding.
* Are able to swallow capsules and tablets.

Exclusion Criteria:

* Have previously completed or withdrawn from this study or any other study investigating LY3039478 or other Notch inhibitors.
* Have evidence of uncontrolled, active infection <7 days prior to administration of study medication.
* Have current or recent gastrointestinal disease with chronic or intermittent diarrhea, or disorders that increase the risk of diarrhea, such as inflammatory bowel disease.
* Have active leukemic involvement of the central nervous system (CNS).

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (22):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University of Texas MD Anderson, Houston, Texas
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Pierre-Bénite
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Toulouse
- Germany (3):
  - Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt
  - Universitätsklinikum Heidelberg, Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Ulm
- Israel (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ramat Gan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Torino

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Borthakur G, Martinelli G, Raffoux E, Chevallier P, Chromik J, Lithio A, Smith CL, Yuen E, Oakley GJ 3rd, Benhadji KA, DeAngelo DJ. Phase 1 study to evaluate Crenigacestat (LY3039478) in combination with dexamethasone in patients with T-cell acute lymphoblastic leukemia and lymphoma. Cancer. 2021 Feb 1;127(3):372-380. doi: 10.1002/cncr.33188. Epub 2020 Oct 27. PMID 33107983
- See also: Click here for more information about this study: A Study of LY3039478 in Combination With Dexamethasone in Participants With T-ALL/T-LBL — http://www.lillytrialguide.com/en-US/studies/leukemia/JJCB#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study completers are those participants that completed Part A cycle 1 or experienced a DLT. There were no participants enrolled to Part B and Phase 2 of the study.
Groups:
- 50 mg LY3039478 + Dexamethasone: Part A: 50 mg LY3039478 administered orally three times per week (TIW) and 24 mg dexamethasone administered orally on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
- 75 mg LY3039478 + Dexamethasone: Part A: 75 mg LY3039478 administered orally three times per week (TIW) and 24 mg dexamethasone administered orally on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
- 100 mg LY3039478 + Dexamethasone: Part A: 100 mg LY3039478 administered orally three times per week (TIW) and 24 mg dexamethasone administered orally on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
- 125 mg LY3039478 + Dexamethasone: Part A: 125 mg LY3039478 administered orally three times per week (TIW) and 24 mg dexamethasone administered orally on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
Period: Overall Study
Arm/Group | 50 mg LY3039478 + Dexamethasone | 75 mg LY3039478 + Dexamethasone | 100 mg LY3039478 + Dexamethasone | 125 mg LY3039478 + Dexamethasone
Started | 6 | 12 | 15 | 3
Completed | 3 | 7 | 11 | 3
Not Completed | 3 | 5 | 4 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Death | 1 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 1 | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 mg LY3039478 + Dexamethasone | 75 mg LY3039478 + Dexamethasone | 100 mg LY3039478 + Dexamethasone | 125 mg LY3039478 + Dexamethasone | Total
Number analyzed (Participants) | 6 | 12 | 15 | 3 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.83 (12.22) | 36.42 (13.40) | 45.87 (14.41) | 26.67 (10.69) | 39.94 (14.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 5 | 1 | 11
  Male | 6 | 7 | 10 | 2 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 4
  Not Hispanic or Latino | 4 | 8 | 11 | 2 | 25
  Unknown or Not Reported | 1 | 3 | 3 | 0 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 5 | 10 | 12 | 3 | 30
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 7 | 7 | 1 | 17
  Italy | 0 | 0 | 2 | 2 | 4
  France | 3 | 4 | 4 | 0 | 11
  Germany | 1 | 1 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT was an Adverse Event(AE) observed during the first 28 day cycle that is determined by the investigator to be at least possibly related to LY3039478 according to CTCAE v 4.0 and fulfills any of the following criteria: CTCAE Grade 3 nonhematological toxicity with a few exceptions, any other significant toxicity deemed to be dose limiting (eg, any toxicity that is possibly related to the study medication that requires the withdrawal of the patient from the study during Cycle 1).
Time Frame: Cycle 1 (Up To 28 Days)
Population: All participants who received at least one dose of study drug in Part A.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg LY3039478 + Dexamethasone | 75 mg LY3039478 + Dexamethasone | 100 mg LY3039478 + Dexamethasone | 125 mg LY3039478 + Dexamethasone
Number analyzed (Participants) | 6 | 12 | 15 | 3
Participants | 0 | 2 | 2 | 3

2. Primary Outcome: Recommended Dose of LY3039478 in Combination With Dexamethasone
Description: A DLT was an Adverse Event(AE) observed during the first 28 day cycle that is determined by the investigator to be at least possibly related to LY3039478 according to CTCAE v 4.0 and fulfills any of the following criteria:CTCAE Grade 3 nonhematological toxicity with a few exceptions, any other significant toxicity deemed to be dose limiting.A dose-limiting equivalent toxicity (DLET) was defined as an AE occurring between Day 1 and Day 28 of any cycle (other than Cycle 1) for a patient enrolled in the Phase 1 portion or in any cycle (including Cycle 1) for a patient enrolled in the Phase 2 portion that would have met the criteria for DLT if it had occurred during Cycle 1 for a patient enrolled in the Phase 1 portion.
Time Frame: Cycle 1 (28 Days)
Population: All participants who received at least one dose of study drug in Part A.
Measure: Number; unit: mg
Groups:
- All Participants: Part A:
  50 mg LY3039478 administered orally three times per week (TIW) and 24 mg dexamethasone administered orally on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
  75 mg LY3039478 administered orally three times per week (TIW) and 24 mg dexamethasone administered orally on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
  100 mg LY3039478 administered orally three times per week (TIW) and 24 mg dexamethasone administered orally on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
  125 mg LY3039478 administered orally three times per week (TIW) and 24 mg dexamethasone administered orally on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
Arm/Group | All Participants
Number analyzed (Participants) | 36
mg | 75

3. Primary Outcome: Number of Participants Who Achieve Complete Remission (CR) or CR With Incomplete Blood Count Recovery (CRi): Overall Remission Rate (ORR)
Description: ORR is defined as the number of participants who achieved a best overall response of either complete remission (CR) or incomplete remission (CRi). The ORR (CR and CRi) is the sum of patients achieving a CR or a CRi divided by the total number of patients randomized in that arm. CR is defined as the number of participants who achieved a best overall response of complete remission (CR), out of the total number of participants randomized in that arm.
Time Frame: Baseline to Objective Disease Progression (Up To 2 Months)
Population: All participants who received at least one dose of study drug in Part A.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg LY3039478 + Dexamethasone | 75 mg LY3039478 + Dexamethasone | 100 mg LY3039478 + Dexamethasone | 125 mg LY3039478 + Dexamethasone
Number analyzed (Participants) | 6 | 12 | 15 | 3
Participants | 1 | 0 | 0 | 0

4. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration-Time Curve (AUC[0-∞]) of LY3039478 in Combination With Dexamethasone in Day 1
Description: Pharmacokinetics (PK): Area Under the Concentration-Time Curve (AUC[0-∞]) of LY3039478 in Combination with Dexamethasone in Day 1
Time Frame: Cycle 1 Day 1: Predose, 1-2, 3-4,6-8,24-30 hours
Population: All participants who received at least one dose of study drug in Part A and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hour per milliliter (ng*h/mL)
Arm/Group | 50 mg LY3039478 + Dexamethasone | 75 mg LY3039478 + Dexamethasone | 100 mg LY3039478 + Dexamethasone | 125 mg LY3039478 + Dexamethasone
Number analyzed (Participants) | 5 | 12 | 15 | 2
nanogram hour per milliliter (ng*h/mL) | 3480 (26) | 5000 (45) | 5870 (49) | 6330 (NA) — For n=2, range 3180-12600 was reported.

5. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration-Time Curve (AUC[0- 48]) of LY3039478 in Combination With Dexamethasone in Day 8
Description: Pharmacokinetics (PK): Area Under the Concentration-Time Curve (AUC[0- 48]) of LY3039478 in Combination with Dexamethasone in Day 8
Time Frame: Cycle 1 Day 8: Predose, 1-2, 3-4,6-8,24-30 hours
Population: All participants who received at least one dose of study drug in Part A and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 50 mg LY3039478 + Dexamethasone | 75 mg LY3039478 + Dexamethasone | 100 mg LY3039478 + Dexamethasone | 125 mg LY3039478 + Dexamethasone
Number analyzed (Participants) | 5 | 8 | 12 | 2
ng*h/mL | 3050 (18) | 4070 (92) | 4640 (55) | 8240 (NA) — For n=2, range 4410-16100 was reported.

6. Secondary Outcome: Number of Participants With CR or CRi and Notch-1 or FBXW7 Mutations
Description: ORR is defined as the number of participants who achieved a best overall response of either complete remission (CR) or incomplete remission (CRi). The ORR (CR and CRi) is the sum of participants achieving a CR or a CRi divided by the total number of participants randomized in that arm. CR is defined as the number of participants who achieved a best overall response of complete remission (CR), out of the total number of participants randomized in that arm.
Time Frame: Baseline to Objective Disease Progression (Up To 12 Months)
Population: All participants who received at least one dose of study drug in Part A.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg LY3039478 + Dexamethasone | 75 mg LY3039478 + Dexamethasone | 100 mg LY3039478 + Dexamethasone | 125 mg LY3039478 + Dexamethasone
Number analyzed (Participants) | 6 | 12 | 15 | 3
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Phase 2: Number of Participants Who Achieve CR, CRi or Partial Remission (PR): Overall Remission Rate (ORR) Plus PR
Time Frame: Baseline to Objective Disease Progression (Up To 12 Months)
Population: Zero participants analyzed. There were no participants enrolled in Phase 2 of the study.
Groups:
- LY3039478 + Dexamethasone: LY3039478 administered orally three times per week (TIW) and 24 mg dexamethasone administered orally on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
- Placebo + Dexamethasone: Placebo administered orally three times per week (TIW) and 24 mg dexamethasone administered orally on days 1-5 every other week during 28 day cycles. Participants receiving benefit may continue until disease progression.
Arm/Group | LY3039478 + Dexamethasone | Placebo + Dexamethasone
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Phase 2: Number of Participants Who Achieve PR
Time Frame: Baseline to Objective Disease Progression (Up To 12 Months)
Population: Zero participants analyzed. There were no participants enrolled in Phase 2 of the study.
Arm/Group | LY3039478 + Dexamethasone | Placebo + Dexamethasone
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Phase 2: Duration of Remission (DoR)
Time Frame: Date of CR, CRi, or PR to Date of Relapse or Death from Any Cause (Approximately 1 Year)
Population: Zero participants analyzed. There were no participants enrolled in Phase 2 of the study.
Arm/Group | LY3039478 + Dexamethasone | Placebo + Dexamethasone
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Phase 2:Relapse Free Survival (RFS)
Time Frame: Date of CR to Relapse or Death from any Cause (Approximately 1 Year)
Population: Zero participants analyzed. There were no participants enrolled in Phase 2 of the study.
Arm/Group | LY3039478 + Dexamethasone | Placebo + Dexamethasone
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Phase 2: Event Free Survival (EFS)
Time Frame: Baseline to Objective Disease Progression or Death from Any Cause (Approximately 1 Year)
Population: Zero participants analyzed. There were no participants enrolled in Phase 2 of the study.
Arm/Group | LY3039478 + Dexamethasone | Placebo + Dexamethasone
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Phase 2: Overall Survival (OS)
Time Frame: Baseline to the Date of Death from Any Cause (Approximately 1.5 Years)
Population: Zero participants analyzed. There were no participants enrolled in Phase 2 of the study.
Arm/Group | LY3039478 + Dexamethasone | Placebo + Dexamethasone
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Phase 2: Change From Baseline in the Functional Assessment of Cancer Therapy-Leukemia-General (FACT-Leu-G) Score
Time Frame: Baseline, End of Study (Approximately 1.5 Years)
Population: Zero participants analyzed. There were no participants enrolled in Phase 2 of the study.
Arm/Group | LY3039478 + Dexamethasone | Placebo + Dexamethasone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up To 16 Months
Arm/Group | 50 mg LY3039478 + Dexamethasone | 75 mg LY3039478 + Dexamethasone | 100 mg LY3039478 + Dexamethasone | 125 mg LY3039478 + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 6/6 | 8/12 | 12/15 | 2/3
Serious Adverse Events (participants affected / at risk) | 6/6 | 11/12 | 9/15 | 3/3
Other Adverse Events (participants affected / at risk) | 6/6 | 12/12 | 15/15 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 mg LY3039478 + Dexamethasone (N=6) | 75 mg LY3039478 + Dexamethasone (N=12) | 100 mg LY3039478 + Dexamethasone (N=15) | 125 mg LY3039478 + Dexamethasone (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 2 (3) | 2 (4) | 1 (5)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
H1n1 influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Neutropenic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (3) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (1) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 mg LY3039478 + Dexamethasone (N=6) | 75 mg LY3039478 + Dexamethasone (N=12) | 100 mg LY3039478 + Dexamethasone (N=15) | 125 mg LY3039478 + Dexamethasone (N=3)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 2 (3) | 3 (4) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exophthalmos (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 7 (20) | 8 (19) | 2 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (8) | 5 (6) | 3 (8)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4) | 8 (8) | 3 (9)
Asthenia (General disorders) | 0 (0) | 3 (5) | 3 (3) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 6 (10) | 2 (8)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 1 (3) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (4) | 4 (4) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatophytosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epstein-barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective glossitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic encephalopathy (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (4) | 3 (5) | 1 (2)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (6) | 4 (8) | 1 (3)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 2 (4) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Blood phosphorus increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 1 (5) | 0 (0)
Chest x-ray abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 1 (5)
Immunoglobulins decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (2) | 2 (8) | 4 (8) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 2 (9) | 0 (0)
Weight decreased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 5 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 5 (7) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (5) | 8 (14) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (8) | 2 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (5)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypouricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dysphoria (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 4 (5) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 6 (6) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 4 (4) | 1 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (3) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
There were no participants enrolled to Part B and Phase 2 of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-06-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT02518113/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT02518113/SAP_001.pdf